CLINICAL TRIAL: NCT07329556
Title: Evaluation of Advanced Glycation End Products Accumulation in Rheumatic Diseases Using Non-Invasive Skin Autofluorescence Measurements
Brief Title: Skin Autofluorescence Assessment of Advanced Glycation End Products in Rheumatic Diseases
Status: Not yet recruiting | Type: Observational
Sponsor: Bursa City Hospital (Other Government)
Responsible Party: Principal Investigator, Taner Dandinoğlu, Principal Investigator, Bursa City Hospital
Other Study IDs: 2026-Rheumatology-1
Record Dates: First submitted 2025-12-28; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Rheumatoid Arthritis (RA; Ankylosing Spondylitis; Psoriatic Arthritis; Reactive Arthritis (ReA); Crystal Arthropathies; Connective Tissue Diseases; Familial Mediterranean Fever (FMF )
MeSH Terms: conditions — Arthritis, Rheumatoid; Spondylitis, Ankylosing; Arthritis, Psoriatic; Arthritis, Reactive; Crystal Arthropathies; Connective Tissue Diseases; Familial Mediterranean Fever

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Rheumatic Diseases Group: Patients diagnosed with inflammatory rheumatic diseases undergoing skin autofluorescence measurement.
- Healthy Control Group: Age- and sex-matched healthy volunteers without a diagnosis of rheumatic disease.

SUMMARY:
Rheumatic diseases are chronic inflammatory conditions that can lead to long-term tissue damage and increased cardiovascular and metabolic risk. Advanced glycation end products (AGEs) are harmful molecules that accumulate in the body over time and are known to promote inflammation and oxidative stress. Increased AGE burden has been implicated in several chronic diseases; however, its role in rheumatic diseases has not been fully clarified.

This observational, cross-sectional study aims to evaluate the accumulation of AGEs in patients with various rheumatic diseases compared with healthy individuals. AGE levels will be assessed non-invasively using skin autofluorescence measurements.

By comparing AGE burden between patients and healthy controls, this study seeks to improve understanding of the potential role of AGEs in the pathophysiology of rheumatic diseases and to explore their usefulness as a non-invasive biomarker in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years
* Diagnosis of an inflammatory rheumatic disease (including rheumatoid arthritis, ankylosing spondylitis, psoriatic arthritis, reactive arthritis, connective tissue diseases, Behçet disease, familial Mediterranean fever, or crystal arthropathies), confirmed by a rheumatologist
* Healthy volunteers without a history of rheumatic or chronic inflammatory disease (for the control group)
* Ability to undergo non-invasive skin autofluorescence measurement
* Ability and willingness to provide written informed consent

Exclusion Criteria:

* Diagnosis of diabetes mellitus (type 1 or type 2)
* Chronic kidney disease with estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73 m²
* Active malignancy or history of malignancy within the past 5 years
* Presence of acute infection or acute inflammatory condition at the time of assessment
* Secondary causes of systemic inflammation unrelated to the underlying rheumatic disease (e.g., uncontrolled endocrine disorders, chronic liver disease)
* Use of medications known to markedly affect AGE accumulation or skin autofluorescence measurements (e.g., recent high-dose systemic glucocorticoids)
* Pregnancy or breastfeeding
* Presence of significant skin conditions (e.g., extensive dermatitis, scars, tattoos, or burns) at the measurement site that may interfere with skin autofluorescence assessment
* Inability to comply with study procedures or to provide informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients aged 18 to 75 years diagnosed with inflammatory rheumatic diseases who are followed at a tertiary rheumatology outpatient clinic, as well as age- and sex-matched healthy volunteers without a history of rheumatic or chronic inflammatory disease. All participants will undergo a single, non-invasive skin autofluorescence measurement to assess advanced glycation end-product (AGE) accumulation.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-04-15 (Estimated)

PRIMARY OUTCOMES:
Skin Autofluorescence-Derived Advanced Glycation End Product Level | Baseline (single study visit)
  Advanced glycation end-product (AGE) accumulation assessed non-invasively by skin autofluorescence measurement using a validated AGE Reader device, expressed in arbitrary units (AU).

SECONDARY OUTCOMES:
Comparison of AGE Levels Between Rheumatic Disease Subtypes | Baseline (single study visit)
  Comparison of skin autofluorescence-derived advanced glycation end-product (AGE) levels among different rheumatic disease subgroups and healthy controls.
Association Between AGE Levels and Inflammatory Markers | Baseline
  Association between skin autofluorescence-derived AGE levels and systemic inflammatory markers, including C-reactive protein (CRP) and erythrocyte sedimentation rate (ESR).

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] de Groot L, Hinkema H, Westra J, Smit AJ, Kallenberg CG, Bijl M, Posthumus MD. Advanced glycation endproducts are increased in rheumatoid arthritis patients with controlled disease. Arthritis Res Ther. 2011;13(6):R205. doi: 10.1186/ar3538. Epub 2011 Dec 14. PMID 22168993